CLINICAL TRIAL: NCT00046449
Title: Prevention of Seasonal Affective Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 398149; NCT00300144 (obsolete NCT alias)
Record Dates: First submitted 2002-09-30; First posted 2002-10-02 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Seasonal Affective Disorder (SAD)
MeSH Terms: conditions — Seasonal Affective Disorder | interventions — Sagittal Abdominal Diameter; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Investigational Seasonal Affective Disorder (SAD) Drug

SUMMARY:
A Placebo Controlled Study Evaluating The Effectivess Of Medication In Preventing Seasonal Affective Disorder

ELIGIBILITY:
Inclusion Criteria: (Patient must meet these criteria in order to be eligible for this study.)

* Patient has a history of Major Depressive Disorder (MDD) with a seasonal pattern.

Exclusion Criteria: (Patient cannot meet these criteria in order to be eligible for this study.)

* Patient has a current or past history of seizure disorder or brain injury.
* Patient has a history or current diagnosis of anorexia nervousa or bulimia.
* Patient has recurrent summer depression more frequently than winter depression.
* Patient has primary diagnosis of panic disorder, Obsessive Compulsive Disorder (OCD), Posttraumatic Stress Disorder (PTSD), acute distress disorder, bipolar II disorder or other psychotic disorders.
* Patient has initiated psychotherapy within the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-09; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (50):
- United States (43):
  - Study Site, Homer, Alaska
  - Study Site, New Haven, Connecticut
  - Study Site, Newark, Delaware
  - Study Site, Wilmington, Delaware
  - Study Site, Washington D.C., District of Columbia
  - Study Site, Boise, Idaho
  - Study SIte, Chicago, Illinois
  - Study Site, Chicago, Illinois
  - Study Site, Hoffman Estates, Illinois
  - Study Site, Libertyville, Illinois
  - Study SIte, Northfield, Illinois
  - Study Site, Schaumburg, Illinois
  - Study SIte, Greenwood, Indiana
  - Study Site, Indianapolis, Indiana
  - Study Site, Florence, Kentucky
  - Study Site, Wellesley Hills, Massachusetts
  - Study Site, Okemos, Michigan
  - Study Site, Royal Oak, Michigan
  - Study Site, Minneapolis, Minnesota
  - Study Site, Moorestown, New Jersey
  - Study Site, Piscataway, New Jersey
  - Study Site, Amityville, New York
  - Study Site, Lawrence, New York
  - Study Site, New York, New York
  - Study Site, Olean, New York
  - Study Site, Staten Island, New York
  - Study Site, Williamsville, New York
  - Study Site, Cincinnati, Ohio
  - Study Site, Cleveland, Ohio
  - Study Site, Independence, Ohio
  - Study Site, Lyndhurst, Ohio
  - Study Site, Toledo, Ohio
  - Study Site, Eugene, Oregon
  - Study Site, Portland, Oregon
  - Study Site, Salem, Oregon
  - Study Site, Allentown, Pennsylvania
  - Study Site, Philadelphia, Pennsylvania
  - Study Site, Lincoln, Rhode Island
  - Study Site, Seattle, Washington
  - Study Site, Madison, Wisconsin
  - Study Site, Middleton, Wisconsin
  - Study Site, Milwaukee, Wisconsin
  - Study Site, West Allis, Wisconsin
- Canada (7):
  - Study Site, Edmonton, Alberta
  - Study Site, Vancouver, British Columbia
  - Study Site, Miramichi, New Brunswick
  - Study Site, Sydney, Nova Scotia
  - Study Site, Markham, Ontario
  - Study Site, Mississauga, Ontario
  - Study Site, Hull, Quebec